CLINICAL TRIAL: NCT06657937
Title: ANKHEAL - Evaluation of the Recovery Experienced by Patients After an Ankle Sprain Treated in the Emergency Department of Nantes University Hospital
Brief Title: Evaluation of the Recovery Experienced by Patients After an Ankle Sprain Treated in the Emergency Department of Nantes University Hospital
Acronym: ANKHEAL
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0524
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Ankle Sprains
Keywords: Emergency; Healing; Ankle; Sprain
MeSH Terms: conditions — Ankle Injuries; Emergencies; Sprains and Strains | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study population: The study population must correspond to the research inclusion criteria:
  Adult patients admitted to the emergency department, presenting with an ankle sprain
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — An initial questionnaire is completed on D0, the day of the patient's admission to the emergency department, by the practitioner in charge of the patient, and covers the patient's anamnesis, clinical examination, radiological examinations and treatment.
  A follow-up telephone visit is then carried out at 30 days by an investigator, to gather information on the clinical and therapeutic evolution, and to evaluate the recovery and evolution of symptoms experienced by the patient in relation to the initial management.
  Other Names: Phone call

SUMMARY:
To evaluate the recovery experienced by patients with ankle sprains treated in the adult emergency department of Nantes University Hospital.

DETAILED DESCRIPTION:
The aim of this study is therefore to establish the current situation by describing the practices of doctors working in the adult emergency department of the Nantes University Hospital regarding the initial treatment of ankle sprains, and to assess the rate of recovery experienced by patients one month after their trauma. This preliminary study may be pursued in the future, with a view to proposing new recommendations for the management of ankle sprains in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Presenting an isolated ankle sprain
* Visiting Nantes CHU emergency department for this reason
* Patient able to read and speak French
* Patient covered by a social security scheme

Exclusion Criteria:

* Patient > 70 years old
* Patients requiring hospitalization following a visit to the emergency department
* Any intercurrent pathology that may affect the management of the ankle sprain
* Associated ankle fracture
* Patients under legal protection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients admitted to adult emergency departments with ankle sprains.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the recovery experienced by patients with ankle sprains treated in the adult emergency department of Nantes University Hospital. | 30 days
  Percentage of patients feeling fully cured at D30

SECONDARY OUTCOMES:
Compare healing sensation with different types of immobilization | 30 days
  Rate of patients feeling fully healed at D30 according to type of immobilization
Compare healing sensation with duration of immobilization | 30 days
  Rate of patients feeling fully healed at D30 according to length of immobilization
Compare the feeling of healing with the initial analgesic proposed | 30 days
  Rate of patients feeling fully healed at D30 according to initial analgesia proposed
Comparing the feeling of recovery according to whether or not a state-certified physiotherapist was involved in the treatment | 30 days
  Rate of patients feeling fully healed at D30 according to whether or not they were treated by a state-qualified physiotherapist
Compare the feeling of recovery according to the presence or absence of early medical reassessment | 30 days
  Rate of patients feeling fully cured at D30 according to the presence or absence of an early medical reassessment
Identify discharge prescription patterns of patients admitted for ankle sprains | 30 days
  Prescription rates for each of the immobilization, analgesia and remote consultation modalities
Identify patients who finally received an alternative diagnosis | 30 days
  Rate of patients receiving an alternative diagnosis
Assessing patients' quality of life at D30 after an ankle sprain | 30 days
  Measurement of median and interquartile range of EQ-5D-5L (EuroQol 5 Dimensions 5 Levels) questionnaire results. The scale ranges from 5 (worst possible health state) to 1 (best possible health state).

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided